CLINICAL TRIAL: NCT06056609
Title: Mother and Baby Yoga Study - Investigating the Influence of an Early Postnatal Mother and Baby Yoga Programme on Maternal Mental Health and Relationship With Baby: a Randomised Feasibility Study.
Brief Title: Mother and Baby Yoga Study - Early Postnatal Yoga and Mental Health
Acronym: MABY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 294028YNP
Record Dates: First submitted 2023-09-05; First posted 2023-09-28 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Issue; Depression, Postpartum; Anxiety
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga - Intervention Group (Active Comparator): The participants in the intervention group (n.20) will obtain access to an eight-week online mother and baby programme. They will be given access to one video per week and asked to complete the session at least once within the week. The participants are also free to repeat the session as many times as they wish.
  The researchers will record the participants access to the online videos. All participants will be asked to complete a daily activity diary.
  The participants will be asked to complete pre, intermediate, and post intervention questionnaires relating to maternal mental health, body satisfaction, and their feelings about the mother and infant bond.
  A subset of participants will also undergo a telephone interview upon completion of the study, which will be subject to qualitative analysis. A short two weekly questionnaire will be sent to all participants for the duration of the study to monitor participant mood and allow for follow up should it be deemed necessary.
  Interventions: Other: Yoga
- Control Group (No Intervention): The participants in the control group (n. 20) will follow the usual standard care pathway and will be offered access to the programme at the end of the study.

INTERVENTIONS:
Other: Yoga — An 8 week online mother and baby yoga programme to include daily diary completion and questionnaires at designated study timepoints
  Arms: Yoga - Intervention Group

SUMMARY:
Investigating the influence of an early postnatal mother and baby yoga programme on maternal mental health and relationship with baby: a randomised feasibility study.

It is thought postnatal mother and baby yoga decreases levels of depression and anxiety and increases subjective experience of maternal-infant bonding. This project will provide the necessary data to determine whether a regular programme would be beneficial to mothers.

The research study is an eight-week online programme incorporating gentle postnatal mother and baby yoga involving women 6-12 weeks following birth (at recruitment/study commencement). The outcome measures include mothers' feelings about their mental health and bond with their baby.

DETAILED DESCRIPTION:
The intended research is an eight-week online programme incorporating gentle postnatal mother and baby yoga.The project will provide essential pilot data to help determine whether mother and baby yoga would be beneficial if offered as a regular service. To achieve this aim, the following study objectives will be addressed:

1. Identify possible links between participation a in programme of mother and baby yoga and maternal subjective experience with mental health
2. Verify whether mother and baby yoga can influence mothers feelings about the bond with their baby
3. Request feedback from the participants to examine the feasibility of running a similar larger study

The outcome measures include mental health and feelings about bonding. The project will provide essential pilot data to help determine whether parent and baby yoga would be acceptable and beneficial if offered as a regular service. Pregnant women and new mothers have suffered negative mental health impacts of COVID-19. An online course has been designed to mitigate anxieties associated with the pandemic, enabling women to follow the course in their own time within a safe environment.

The mental health of women during and after pregnancy is of major concern to health professionals, families and society. 20% of women develop mental health problems during pregnancy or within a year of giving birth. Mental health is the third largest cause of direct maternal deaths during or within 42 days of pregnancy. Suicide is the leading cause of maternal death within a year of giving birth.

Perinatal mental health problems in the UK cost £8.1 billion per year. The average cost to society of one case of perinatal depression is around £74,000, of which £23,000 relates to the mother and £51,000 relates to the impacts on the child. The cost of mental health to the public sector is five times more than the cost of improving mental health services.

Improving outcomes for women will minimise the negative effects on the infant. NICE add that a woman's ability to provide nurturing depends on her own emotional well-being. The charity Best Beginnings believes that all children regardless of income or background should have the best possible start in life, laying foundations for better future life chances. UNICEF Baby Friendly initiative encourages frequent touch and sensitive communication as this trigger's oxytocin, which facilities babies brain development.

Postnatal mum and baby yoga are two distinct areas of therapy, but work well when practiced together. Current evidence supporting yoga in the perinatal period is limited and mostly focuses on pregnancy. Sheffield and Woods-Giscombé call for more larger studies to validate and extend existing findings that demonstrate the potential of yoga for improving mental health for women and infants.

A systematic review concluded Yoga-based interventions may offer a promising potential intervention for maternal mental health and well-being. However, due to the limited number of studies, and a lack of consistency in study design and measures, more high-quality research is required to establish these effects, assess potential benefits on other aspects of maternal well-being and explore potential benefits for outcomes relating to the infant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* 6-12 weeks post birth or 11-12 weeks if birthed by caesarean section
* Uncomplicated postnatal recovery for mother and infant
* Attended postnatal check with and supported to take part in the study by their GP.
* Understand written and/or spoken English

Exclusion Criteria:

* Age 18 and above
* Under 6 weeks post birth or over 12 weeks post birth
* Under 11 weeks or over 12 weeks if birthed by caesarean
* Not attended postnatal check with GP
* Uncontrolled or new medical condition that will increase the risk of unsupervised exercise (cardiac, musculoskeletal, neurological)
* Recent surgical intervention and still in the recovery period
* Uncontrolled or new treatment for depression and/or anxiety
* Currently recovering from a pregnancy or birth related problem that requires health practitioner follow up (medical, surgical, mental health)
* Neonatal complications (prematurity, birth complications, medical/surgical problems, genetic disorders)
* Drug or alcohol dependency
* Multiple birth
* Unable to understand written and/or spoken English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All eligible participants must be assigned female at birth
Enrollment: 34 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal subjective experience of their mental health during and post online yoga programme | 8 weeks
  This is an explorative feasibility study which will expand current knowledge on the link between participation in a mother and baby yoga program & maternal subjective experience with mental health. Mental health related outcomes are measured using the Edinburgh Postnatal Scale (scores of 10 or more are suggestive of depression requiring further evaluation). Using well-established scales allows for comparison with other studies. A short two weekly questionnaire is sent to all participants for the duration of the study. Many studies have found the Positive Affect Negative Affect Scale (scores range from 10 - 50 on both scales with higher scores on the positive affect scale representing higher levels of positive affect, and lower scores on the negative affect scale representing lower levels of negative affect) to be a reliable and valid tool.
Maternal subjective experience of their mental health during and post online yoga | 8 weeks
  This is an explorative feasibility study which will expand current knowledge on the link between participation in a mother and baby yoga program & maternal subjective experience with mental health. Mental health related outcomes are measured using the Postpartum Specific Anxiety Scale (a score of >112 requires further evaluation). Using well-established scales allows for comparison with other studies. A short two weekly questionnaire is sent to all participants for the duration of the study. Many studies have found the Positive Affect Negative Affect Scale (scores range from 10 - 50 on both scales with higher scores on the positive affect scale representing higher levels of positive affect, and lower scores on the negative affect scale representing lower levels of negative affect) to be a reliable and valid tool.

SECONDARY OUTCOMES:
Maternal subjective feelings and experience towards the body and bond with infant post partum, during and post online yoga programme | 8 weeks
  Secondary outcome measures include feelings towards the body and mother's bond with infant. Feelings toward the body will be measured by the Postpartum Mind and Body scale (PMB). The PMB is 41-item scale with responses made on a 5-point likert scale (ranging from strongly agree to strongly disagree). Body satisfaction is important during the perinatal period in predicting outcomes such as depression and anxiety. Body satisfaction has also been found to relate to antenatal attachment in pregnant samples. Mother and infant bonding will be measured with the Postpartum Bonding Questionnaire. The PBQ is a 25-item measure of parent infant bonding. Responses are made on a 6-point Likert scale ranging from 0 - 5 (0 = always, 5 = never). The scale consists of four subscales: 1) weakened bonding, 2) rejection and pathological rage, 3) anxiety about the baby/anxiety about caring for the baby, and 4) risk of abuse to the baby (the subscale examining risk of abuse will be omitted from this study).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Phillips, Study Chair — York & Scarborough Teaching Hospitals NHS Foundation Trust
Locations (1):
- York & Scarborough Teaching Hospitals NHS Foundation Trust, York, N. Yorks, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durankus F, Aksu E. Effects of the COVID-19 pandemic on anxiety and depressive symptoms in pregnant women: a preliminary study. J Matern Fetal Neonatal Med. 2022 Jan;35(2):205-211. doi: 10.1080/14767058.2020.1763946. Epub 2020 May 18. PMID 32419558
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] Cox JL, Chapman G, Murray D, Jones P. Validation of the Edinburgh Postnatal Depression Scale (EPDS) in non-postnatal women. J Affect Disord. 1996 Jul 29;39(3):185-9. doi: 10.1016/0165-0327(96)00008-0. PMID 8856422
- [Background] Doran F, Hornibrook J. Women's experiences of participation in a pregnancy and postnatal group incorporating yoga and facilitated group discussion: a qualitative evaluation. Women Birth. 2013 Mar;26(1):82-6. doi: 10.1016/j.wombi.2012.06.001. Epub 2012 Jul 19. PMID 22818031
- [Background] Fallon V, Halford JCG, Bennett KM, Harrold JA. The Postpartum Specific Anxiety Scale: development and preliminary validation. Arch Womens Ment Health. 2016 Dec;19(6):1079-1090. doi: 10.1007/s00737-016-0658-9. Epub 2016 Aug 29. PMID 27571782
- [Background] Jiang Q, Wu Z, Zhou L, Dunlop J, Chen P. Effects of yoga intervention during pregnancy: a review for current status. Am J Perinatol. 2015 May;32(6):503-14. doi: 10.1055/s-0034-1396701. Epub 2014 Dec 23. PMID 25535930
- [Background] MacDonald C. Mother and baby yoga is good for you. Pract Midwife. 2013 May;16(5):14, 16, 18. PMID 23789249
- [Background] Sheffield KM, Woods-Giscombe CL. Efficacy, Feasibility, and Acceptability of Perinatal Yoga on Women's Mental Health and Well-Being: A Systematic Literature Review. J Holist Nurs. 2016 Mar;34(1):64-79. doi: 10.1177/0898010115577976. Epub 2015 Apr 20. PMID 25896571
- [Background] Timlin D, Simpson EE. A preliminary randomised control trial of the effects of Dru yoga on psychological well-being in Northern Irish first time mothers. Midwifery. 2017 Mar;46:29-36. doi: 10.1016/j.midw.2017.01.005. Epub 2017 Jan 13. PMID 28129548
- [Background] Vogel L. Tailored treatment for postpartum depression. CMAJ. 2011 Nov 8;183(16):E1163-4. doi: 10.1503/cmaj.109-4003. Epub 2011 Oct 3. No abstract available. PMID 21969408
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- See also: London: Best Beginnings [updated 2020 August 06, cited 2020 August 06]; — https://www.bestbeginnings.org.uk
- See also: Knight M, Bunch K, Tuffnell D, Jayakody H, Shakespeare J, Kotnis R et al. Saving Lives, Improving Mothers' Care: Lessons learned to inform maternity care from the UK and Ireland Confidential Enquiries into Maternal Deaths and Morbidity 2014-16 — https://www.npeu.ox.ac.uk
- See also: NHS England, Improvement NHS, for Mental Health NCC, Others. Implementing the Mental Health Forward View. London: NHS England [Internet] 2017 — https://www.england.nhs.uk/mental-health/taskforce/imp
- See also: National Institute for Health and Care Excellence (NICE). Postnatal care. Quality standard (QS37). London: NICE. [updated: 01 2015 June, cited 2020 August]; — https://www.nice.org.uk/guidance/qs37
- See also: Preston, C. & Kirk, E (2020 December 16th). Postnatal Mind and Body. [Webinar Presentation]. Becoming Mothers: Perinatal Mind and Body Research - Postnatal Bodies. University of York UK — https://youtu.be/ZtVVHRzYy4A
- See also: Royal College of Psychiatrists. COVID-19: Mental health before, during and after pregnancy [Internet]. London: Royal College of Psychiatrists [updated 2020 August 01, cited 2020 August 06] — https://www.rcpsych.ac.uk/mental-health/treatments-and-wellbeing/perinatal-care-and-covid-19
- See also: The Baby Friendly Initiative. Building a Happy Baby A Guide for Parents [Internet]; London: UNICEF UK [updated 2019 March, cited 2020 August]. — https://www.unicef.org.uk/babyfriendly/wp-content/uploads/sites/2/2018/04/happybaby_leaflet_web.pdf